CLINICAL TRIAL: NCT05125757
Title: Response of Fatty Liver to Lifestyle Modification in Psoriasis Patients
Brief Title: Lifestyle Modification in Psoriatic Patients With Fatty Liver
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003344
Record Dates: First submitted 2021-10-17; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Psoriasis; Fatty Liver
MeSH Terms: conditions — Psoriasis; Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): The patients of this group will receive their usual immuno-modulating therapy plus life style modification (energy or diet restriction in addition to daily walking, 15000 steps)
  Interventions: Other: lifestyle modification
- control group (Active Comparator): The participants of this group will receive their usual immuno-modulating therapy and continuing their usual diet and activities
  Interventions: Other: usual lifestyle

INTERVENTIONS:
Other: lifestyle modification — for 12 week, the patients of this group will receive their usual immuno-modulating therapy plus life style modification (energy or diet restriction in addition to daily walking, 15000 steps)
  Arms: intervention group
Other: usual lifestyle — the patients will receive the usual immuno-modulating therapy with continued usual diet and activities
  Arms: control group

SUMMARY:
Several recent reports have shown an increased prevalence of nonalcoholic fatty liver disease (NAFLD) in those with psoriasis, which may reflect the increased occurrence of metabolic syndrome in this patient population.

DETAILED DESCRIPTION:
the recruitment of 60 fatty live men with chronic disease, psoriasis, will be classified to lifestyle modification group (foe 12 weeks, this patients will take supervised energy or diet restriction program plus their usual immunosuppressive drugs ) and control group will continue their drug program only)

ELIGIBILITY:
Inclusion Criteria:

* psoriasis obese patients with coexisting fatty liver
* chronic plaque psoriasis
* patients who will not show any change in immuno-modulating psoriasis therapies for at least five months before participation in the study.

Exclusion Criteria:

* no metabolic syndrome
* no renal or cardiac or pulmonary disorders
* other types of psoriasis

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation of gender identity
Enrollment: 60 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index | It will be measured after 12 weeks
  it is an index used to measure level and severity of psoriasis

SECONDARY OUTCOMES:
Dermatology Life Quality Index | It will be measured after 12 weeks
  it is a questinnaire used to assess life quality in psoriasis humans
triglycerides | It will be measured after 12 weeks
  will measured in plasma
AST | It will be measured after 12 weeks
  it is plasma aspartate transaminase
ALT | It will be measured after 12 weeks
  it is plasma Alanine transaminase
BMI | It will be measured after 12 weeks
  it is body mass index
waist circumference | It will be measured after 12 weeks
  it will be measured at the level of umbilicus

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Dokki, Egypt